CLINICAL TRIAL: NCT02549300
Title: Konnektif Doku Masajı ve Yaşam Stili Modifikasyonlarının Adölesanlarda Gerilim Tipi Baş Ağrısına Etkisi
Brief Title: The Effects of Connective Tissue Massage and Lifestyle Modifications in Adolescents Tension Type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emine BARAN, Research Assistant Emine Baran, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU
Record Dates: First submitted 2015-03-18; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Headache Disorders, Primary
Keywords: connective tissue massage; adolescent tension-type headache
MeSH Terms: conditions — Headache Disorders, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): 15 patients will be included in control group. Control group will just receive advices about life style modifications, such as teaching good postural habits, using right glasses, not smoking, regular and quality sleep habits.
- Study Group (Experimental): 15 patients will be included in study group. Study group will be treated with connective tissue massage in addition to life style modifications (such as teaching good postural habits, using right glasses, not smoking, regular and quality sleep habits.). Connective tissue massage will be applied 5 times a week, totally 20 sessions in a month. Each session lasts approximately 20-30 minutes. Connective tissue massage will be applied on basic part, lower thoracic, scapular, inter scapular and neck regions.
  Interventions: Other: Connective tissue massage

INTERVENTIONS:
Other: Connective tissue massage — It is a manual reflex therapy in that it is applied with the therapist's hands which are in contact with the patient's skin. The assessment of the patient and the clinical decision-making that directs treatment is based on a theoretical model that assumes a reflex effect on the autonomic nervous system which is induced by manipulating the fascial layers within and beneath the skin.
  Other Names: connective tissue manipulation
  Arms: Study Group

SUMMARY:
The purpose of this study is to investigate the effects of connective tissue massage and lifestyle modifications in adolescents tension type headache, pain severity, pain duration, pain frequency and quality of life and pressure pain threshold rates. The patients will be accepted to study according to 'The International Classification of Headache Disorders-III' criteria. Including criteria are; being between 10-19 ages adolescents, suffering from tension type headache at least for 6 months, pain severity between 4-7 on visual analog scale. Excluding criteria are; current pregnancy, having any history of cancer, traffic accident, head trauma and any kind of neurological disorder. Patients will be divided into two groups randomly. The investigators plan to receive 30 patients to the study. 15 of them will be in control group, 15 in study group. Control group will just receive some advices including life style modifications, like using right glasses, not smoking, true posture habits and regular and quality sleep habits. In addition to life style modifications, the other group will be treated with connective tissue massage. Connective tissue massage will be applied on basic part, lower thoracic, scapular, inter scapular and neck regions, 5 times a week, totally 20 sessions in a month. Each session lasts approximately 20-30 minutes. Patients detailed medical history and demographic data will be recorded. Pain severity, duration, frequency, analgesic usage, connective tissue evaluation of back, range of motion of neck, pressure pain threshold for pain sensitization measurements and quality of life will be evaluated before treatment and after 4 weeks of treatment.

DETAILED DESCRIPTION:
The patients will be accepted to study according to 'The International Classification of Headache Disorders-III'. Including criteria are; being between 10-19 aged adolescents, suffering from tension type headache at least for 6 months, pain severity between 4-7 on visual analog scale. Excluding criteria are; current pregnancy, having any history of cancer, traffic accident, head trauma and any kind of neurological disorder. Patients will be divided into two groups randomly. Control group will be taught some advices about life style modifications, like using right glasses, teaching true posture, regular and quality sleep habits. In addition to life style modifications, the other group will be treated with connective tissue massage. Connective tissue massage will be applied 5 times a week, totally 20 sessions in a month. Each session lasts approximately 20-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 10-19 ages
* Prognosed with tension type headache according to 'The International Classification of Headache Disorders-III' criteria
* Suffering from tension type headache for at least 6 months
* Pain severity must be between 4-7 on visual analog scale

Exclusion Criteria:

* Current pregnancy
* Any kind of cancer history
* History of head trauma
* Any kind of neurological disorder
* Receiving physiotherapy in last 6 months
* Unwillingness to participate in the study

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | Change from baseline in pain severity at four weeks
  Pain severity will be measured with McGill Short Form Pain Questionnaire

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (Turkish version of the questionnaire) | Change from baseline in questionnaire at four weeks
Range of motion | Change from baseline in range of motion at four weeks
  Cervical range of motion will be measured with an inclinometer.
Pressure pain threshold | Change from baseline in pressure pain threshold measurement at four weeks
  Pressure pain thresholds will be measured at the dorsum of the second finger (middle phalanx) and at the anterior part of the temporal muscle, where palpation had revealed it to be most prominent.

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Akbayrak, Prof.Dr., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Samanpazarı, Turkey (Türkiye)

REFERENCES:
- [Result] Grimmer K, Nyland L, Milanese S. Repeated measures of recent headache, neck and upper back pain in Australian adolescents. Cephalalgia. 2006 Jul;26(7):843-51. doi: 10.1111/j.1468-2982.2006.01120.x. PMID 16776700
- [Result] Albers L, Milde-Busch A, Bayer O, Lehmann S, Riedel C, Bonfert M, Heinen F, Straube A, von Kries R. Prevention of headache in adolescents: population-attributable risk fraction for risk factors amenable to intervention. Neuropediatrics. 2013 Feb;44(1):40-5. doi: 10.1055/s-0032-1332742. Epub 2013 Jan 8. PMID 23299655
- [Result] Breuner CC, Smith MS, Womack WM. Factors related to school absenteeism in adolescents with recurrent headache. Headache. 2004 Mar;44(3):217-22. doi: 10.1111/j.1526-4610.2004.04050.x. PMID 15012658
- [Result] Oksanen A, Metsahonkala L, Viander S, Jappila E, Aromaa M, Anttila P, Salminen J, Sillanpaa M. Strength and mobility of the neck-shoulder region in adolescent headache. Physiother Theory Pract. 2006 Sep;22(4):163-74. doi: 10.1080/09593980600822800. PMID 16920676
- [Result] Borusiak P, Biedermann H, Bosserhoff S, Opp J. Lack of efficacy of manual therapy in children and adolescents with suspected cervicogenic headache: results of a prospective, randomized, placebo-controlled, and blinded trial. Headache. 2010 Feb;50(2):224-30. doi: 10.1111/j.1526-4610.2009.01550.x. Epub 2009 Oct 21. PMID 19845788
- [Result] Walter S. Lifestyle behaviors and illness-related factors as predictors of recurrent headache in U.S. adolescents. J Neurosci Nurs. 2014 Dec;46(6):337-50. doi: 10.1097/JNN.0000000000000095. PMID 25365048
- [Result] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158
- [Result] Castien RF, van der Windt DA, Grooten A, Dekker J. Effectiveness of manual therapy for chronic tension-type headache: a pragmatic, randomised, clinical trial. Cephalalgia. 2011 Jan;31(2):133-43. doi: 10.1177/0333102410377362. Epub 2010 Jul 20. PMID 20647241
- [Result] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Result] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Result] Olesen J. ICHD-3 beta is published. Use it immediately. Cephalalgia. 2013 Jul;33(9):627-8. doi: 10.1177/0333102413487610. No abstract available. PMID 23771275
- [Result] Buchgreitz L, Lyngberg AC, Bendtsen L, Jensen R. Frequency of headache is related to sensitization: a population study. Pain. 2006 Jul;123(1-2):19-27. doi: 10.1016/j.pain.2006.01.040. Epub 2006 Apr 13. PMID 16630694